CLINICAL TRIAL: NCT03611361
Title: Wound Imaging System to Gather Clinical References: Collection of Clinical References Images for the Second Generation DeepView Wound Imaging System
Brief Title: Wound Imaging Study to Gather Clinical References for a Device to Assist Selecting Level-of-amputation in PAD Patients
Acronym: WISCR
Status: Terminated | Type: Observational
Why Stopped: Able to reach conclusions about feasibility with number of subjects enrolled.
Sponsor: SpectralMD (Industry)
Collaborators: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CP-16-002
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Amputation Wound; Peripheral Arterial Disease
Keywords: peripheral arterial disease; re-amputation; optical imaging; Computer Assisted Detection (CADe)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin punch biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: SpectralMD DeepView Wound Imaging System 2.0 — The DeepView is an imaging device which simultaneously performs multispectral imaging (MSI) measurements across the visible and infrared spectrum to obtain a quantitative tissue viability assessment. These optical measurements are integrated using a machine learning (ML) algorithm to categorize microvascular blood flow and provide a quantitative assessment for selection of tissue healing.

SUMMARY:
This is a proof-of-concept study to collect images to train a CADe algorithm to predict the correct level of amputation in individuals scheduled for amputation secondary to PAD.

DETAILED DESCRIPTION:
SpectralMD has developed an imaging device (DeepView), which simultaneously performs multispectral imaging (MSI) measurements across the visible and infrared spectrum to obtain a quantitative tissue viability assessment. These optical measurements are integrated using a CADe algorithm to categorize microvascular blood flow and provide a quantitative assessment to aid in selecting the appropriate amputation site.

The investigators intend to gather data to train the CADe algorithm to predict ultimate healing status of tissue in the lower extremities of individuals suffering from peripheral arterial disease (PAD). The investigators will demonstrate the feasibility of using such an algorithm to accurately predict the location and extent of small vessel disease prior to amputation. Eventually, the invesitgators expect the DeepView to reduce the rate of re-amputation in patients with peripheral arterial disease if used for routine assessment of patients prior to amputation.

The aims of the study are as follows:

* Evaluate performance of a Computer Assisted Detection (CADe) algorithm trained to assist selecting the level-of-amputation in patients with PAD.
* Identify multispectral signatures that are strongly predictive of viable skin tissue at proposed amputation sites.
* Create a representative database for training the CADe algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Patient must require amputation on a limb secondary to PAD, defined as arterial insufficiency due to atherosclerosis based on one or more of the following assessments:

  * Ankle brachial index;
  * Duplex ultrasonography showing clinically significant occlusion;
  * Arteriography; or
  * Assessment demonstrating stenosis by arterial calcification.
* Able to give informed consent,
* Be at least 18 years of age.

Exclusion Criteria:

* No history of major amputation on the affected limb, or
* Life expectancy less than 6 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with peripheral arterial disease in a lower extremity.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Standardized amputation healing assessment | 30-days
  Healing as indicated by: re-epithelialization of tissue within the incision site and no signs of drainage/exudate.

SECONDARY OUTCOMES:
Standardized amputation healing assessment | 90-days
  Healing as indicated by: re-epithelialization of tissue within the incision site and no signs of drainage/exudate.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Gable, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Dr. Dennis Gable, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kono Y, Muder RR. Identifying the incidence of and risk factors for reamputation among patients who underwent foot amputation. Ann Vasc Surg. 2012 Nov;26(8):1120-6. doi: 10.1016/j.avsg.2012.02.011. Epub 2012 Jul 25. PMID 22840342
- [Background] Zonios G, Bykowski J, Kollias N. Skin melanin, hemoglobin, and light scattering properties can be quantitatively assessed in vivo using diffuse reflectance spectroscopy. J Invest Dermatol. 2001 Dec;117(6):1452-7. doi: 10.1046/j.0022-202x.2001.01577.x. PMID 11886508
- [Background] Thatcher JE, Li W, Rodriguez-Vaqueiro Y, Squiers JJ, Mo W, Lu Y, Plant KD, Sellke E, King DR, Fan W, Martinez-Lorenzo JA, DiMaio JM. Multispectral and Photoplethysmography Optical Imaging Techniques Identify Important Tissue Characteristics in an Animal Model of Tangential Burn Excision. J Burn Care Res. 2016 Jan-Feb;37(1):38-52. doi: 10.1097/BCR.0000000000000317. PMID 26594863